CLINICAL TRIAL: NCT02367404
Title: A Prospective Randomized Controlled Study Comparing the Efficacy of Pelvic Floor Muscle Training and Oral Duloxetine in the Recovery of Continence After Robotic Assisted Radical Prostatectomy
Brief Title: Prospective RCT on Post Prostatectomy Urine Leak
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Mutualiste Montsouris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URO-01-2014
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Prostate Cancer; Urinary Incontinence
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (No Intervention): Keigel's exercise
- Duloxetine (Active Comparator): Duloxetine 60mg for 3 months
  Interventions: Drug: Duloxetine
- Duloxetine + PMFT (Active Comparator): Duloxetine 60mg for 3 months PMFT weekly for 3 months
  Interventions: Drug: Duloxetine; Behavioral: Pelvic Floor Muscle Training
- Pelvic Floor Muscle Training (Active Comparator): PMFT weekly for 3 months
  Interventions: Behavioral: Pelvic Floor Muscle Training

INTERVENTIONS:
Drug: Duloxetine — Duloxetine 60mg OD for 3 months
  Other Names: Cymbalta
  Arms: Duloxetine; Duloxetine + PMFT
Behavioral: Pelvic Floor Muscle Training — PMFT weekly for 3 months
  Other Names: Pelvic Physiotherqpy
  Arms: Duloxetine + PMFT; Pelvic Floor Muscle Training

SUMMARY:
Objectives:

Primary: Comparison of proportion of patient achieving continence between the four arms at 6 months.

Secondary:

* Comparison of time to achieve continence between the four arms.
* Comparison of urinary symptoms and quality of life improvement between the four arms.
* Assessment of adverse events in Duloxetine arms.

Primary outcome/ time frame: Proportion of patient achieving continence at 6 months. Continence is defined as "using no pad"or "only security pad".

Secondary outcome:

* time to achieve continence
* Quality of life tested in relation to incontinence according to Visual Analog Scale (VAS) and King's Health Questionnaire (KQH).
* Urinary symptoms measured with International Prostate Symptom Score (IPSS).

No. of subjects entered: 300 patients informed and included, 240 patients will be randomized.

Statistical methods

* Proportion of patients who achieve continence and time to achieve continence will be compared between the four arms.
* Comparison of quality of life outcomes between the four arms
* Comparison of clinical variables that can affect the primary/secondary outcome - univariate and multivariate analysis (ITT).

ELIGIBILITY:
Inclusion Criteria:

1. All consecutive patients undergoing Robotic Assisted Radical Prostatectomy for clinically organ confined prostate cancer

Exclusion Criteria:

1. Prior urethral, bladder or prostate surgery
2. Pelvic radiotherapy.
3. Overactive bladder
4. Known neurological disease associated to LUTS
5. Hepatic impairment with hepatic insufficiency.
6. Severe renal impairment (creatinine clearance < 30ml/min)
7. Hypersensitivity to duloxetine
8. Uncontrolled hypertension
9. Narrow angle glaucoma

   Post-operative criteria:
10. Post-void residual urine volume > 100ml measured 15 days after the RARP

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-02 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Urinary continence proportion | 6 months
  Proportion of patient achieving continence at 6 months

SECONDARY OUTCOMES:
Urinary continence time | 6 months
  time to achieve continence
Urinary quality of life | 6 months
  Quality of life tested in relation to incontinence using questionnaire at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Sanchez-Salas, MD, Principal Investigator — Institute Mutualiste Montsouris
Locations (1):
- Institut Mutualiste montsouris, Paris, France